CLINICAL TRIAL: NCT03789838
Title: Prospective Cohort Study Examining the Effect of a Sepsis Rapid Response Team in the Emergency Department
Brief Title: Effect of Sepsis Response Team in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Aleksander Rygh Holten, Consultant Physician, Oslo University Hospital
Other Study IDs: Ulleval sepsis-01
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before of sepsis rapid response team: Time from arrival at the Emergency Department to antibiotic is administered, before introduction of sepsis response team in the Emergency Department.
- Sepsis rapid response team: Time from arrival at the Emergency Department to antibiotic is administered, with sepsis response team in the Emergency Department.
  Interventions: Other: Sepsis rapid response team

INTERVENTIONS:
Other: Sepsis rapid response team — Patients with suspected sepsis is managed by a sepsis rapid response team in a structured manner.
  Groups: Sepsis rapid response team

SUMMARY:
Does sepsis response team in the emergency department increase the portion of sepsis patient who receive adequate treatment within one hour?

DETAILED DESCRIPTION:
Does sepsis response team in the emergency department increase the portion of sepsis patient who receive adequate treatment within one hour? The time from the patients arrive at the emergency department to an adequate antibiotic is given, before and after introduction of a sepsis response team, was registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected sepsis

Exclusion Criteria:

* Patients who was consider not to need antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected sepsis in emergency department
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Time from arrival the emergency department to antibiotic is given. | 6 months
  Time from arrival the emergency department to antibiotic is given.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Holten, Phd, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trydal E, Martinsen AB, Beisland F, Jacobsen D, Holten AR. [Structured evaluation on arrival of patients with sepsis and initiation of antibiotics]. Tidsskr Nor Laegeforen. 2019 May 27;139(9). doi: 10.4045/tidsskr.18.0216. Print 2019 May 28. Norwegian. PMID 31140244